CLINICAL TRIAL: NCT03397121
Title: Placebo-Controlled, Double-Blind, Randomized Trial to Evaluate the Effect of 300 mg of Inclisiran Sodium Given as Subcutaneous Injections in Subjects With Heterozygous Familial Hypercholesterolemia (HeFH) and Elevated Low-Density Lipoprotein Cholesterol (LDL-C).
Brief Title: Trial to Evaluate the Effect of Inclisiran Treatment on Low Density Lipoprotein Cholesterol (LDL-C) in Subjects With Heterozygous Familial Hypercholesterolemia (HeFH)
Acronym: ORION-9
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Medicines Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MDCO-PCS-17-03; 2017-002472-30 (EudraCT Number)
Record Dates: First submitted 2018-01-02; First posted 2018-01-11 (Actual); Results first posted 2020-10-28 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Heterozygous Familial Hypercholesterolemia; Elevated Cholesterol
Keywords: HeFH; LDL-C; Inclisiran
MeSH Terms: conditions — Hypercholesterolemia | interventions — ALN-PCS; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Inclisiran (Experimental): Inclisiran sodium 300 milligrams (mg) will be administered as a SC injection on Day 1, Day 90 then every 6 months.
  Interventions: Drug: Inclisiran
- Placebo (Placebo Comparator): Placebo will be administered as SC injections of saline solution on Day 1, Day 90 then every 6 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Inclisiran — Inclisiran is a small interfering ribonucleic acid (RNA) that inhibits PCSK9 synthesis.
  Arms: Inclisiran
Drug: Placebo — Placebo will be supplied as sterile normal saline (0.9% sodium chloride in water for injection).
  Other Names: Saline Solution
  Arms: Placebo

SUMMARY:
This is a Phase III, placebo-controlled, double-blind, randomized study in participants with HeFH and elevated LDL-C to evaluate the efficacy, safety, and tolerability of subcutaneous (SC) injection(s) of inclisiran. The study will be multicenter and international.

ELIGIBILITY:
Inclusion Criteria:

Participants may be included if they meet all of the following inclusion criteria prior to randomization:

1. Male or female participants ≥18 years of age.
2. History of HeFH with a diagnosis of HeFH by genetic testing; and/or a documented history of untreated LDL-C of >190 mg/dL, and a family history of familial hypercholesterolemia, elevated cholesterol or early heart disease that may indicate familial hypercholesterolemia.
3. Serum LDL-C ≥2.6 millimoles (mmol)/liter (L) (≥100 mg/dL) at screening.
4. Fasting triglyceride <4.52 mmol/L (<400 mg/dL) at screening.
5. Participants on statins should be receiving a maximally tolerated dose.
6. Participants not receiving statins must have documented evidence of intolerance to all doses of at least 2 different statins.
7. Participants on lipid-lowering therapies (such as a statin and/or ezetimibe) should be on a stable dose for ≥30 days before screening with no planned medication or dose change during study participation.

Exclusion Criteria:

Participants will be excluded from the study if any of the following exclusion criteria apply immediately prior to randomization:

1. New York Heart Association (NYHA) class IV heart failure.
2. Uncontrolled cardiac arrhythmia
3. Uncontrolled severe hypertension
4. Active liver disease
5. Females who are pregnant or nursing, or who are of childbearing potential and unwilling to use at least 2 methods of highly effective contraception (failure rate less than 1% per year) (combined oral contraceptives, barrier methods, approved contraceptive implant, long-term injectable contraception, or intrauterine device) for the entire duration of the study. Exemptions from this criterion:

   1. Women >2 years postmenopausal (defined as 1 year or longer since last menstrual period) AND more than 55 years of age.
   2. Postmenopausal women (as defined above) and less than 55 years of age with a negative pregnancy test within 24 hours of randomization.
   3. Women who are surgically sterilized at least 3 months prior to enrollment.
6. Males who are unwilling to use an acceptable method of birth control during the entire study period (condom with spermicide).
7. Treatment with other investigational products or devices within 30 days or 5 half-lives of the screening visit, whichever is longer.
8. Treatment (within 90 days of screening) with monoclonal antibodies directed towards PCSK9.

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 482 (Actual)
Dates: Start 2017-11-28 (Actual); Primary Completion 2019-08-27 (Actual); Study Completion 2019-09-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frederick J. Raal, MD, Principal Investigator — University of Witwatersrand, South Africa
Locations (45):
- United States (10):
  - Site 90001-005, Mission Viejo, California
  - Site 90001-001, Newport Beach, California
  - Site 90001-015, Stanford, California
  - Site 90001-047, Boca Raton, Florida
  - Site 90001-004, Boston, Massachusetts
  - Site 90001-056, Saint Paul, Minnesota
  - Site 90001-012, Butte, Montana
  - Site 90001-112, Las Vegas, Nevada
  - Site 90001-014, Summit, New Jersey
  - Site 90001-002, Cincinnati, Ohio
- Canada (3):
  - Site 90011-005, Chicoutimi, Quebec
  - Site 90011-001, Montreal, Quebec
  - Site 90011-002, Québec, Quebec
- Czechia (3):
  - Site 90420-001, Prague
  - Site 90420-006, Prague
  - Site 90420-005, Trutnov
- Denmark (6):
  - Site 90045-001, Aalborg
  - Site 90045-004, Esbjerg
  - Site 90045-003, Herning
  - Site 90045-006, Hvidovre
  - Site 90045-002, Roskilde
  - Site 90045-005, Viborg
- Netherlands (5):
  - Site 90031-001, Amersfoort
  - Site 90031-003, Amsterdam
  - Site 90031-009, Hoorn
  - Site 90031-006, Tilburg
  - Site 90031-005, Utrecht
- South Africa (9):
  - Site 90027-004, Cape Town, Western Cape
  - Site 90027-003, Bloemfontein
  - Site 90027-005, Cape Town
  - Site 90027-001, Cape Town
  - Site 90027-008, Cape Town
  - Site 90027-010, Johannesburg
  - Site 90027-007, Pretoria
  - Site 90027-006, Pretoria
  - Site 90027-009, Witbank
- Spain (6):
  - Site 90034-003, A Coruña
  - Site 90034-005, Barcelona
  - Site 90034-004, Córdoba
  - Site 90034-006, L'Hospitalet de Llobregat
  - Site 90034-001, Reus
  - Site 90034-002, Zaragoza
- Sweden (3):
  - Site 90046-002, Gothenburg
  - Site 90046-001, Stockholm
  - Site 90046-003, Stockholm

REFERENCES:
- [Derived] Dutta S, Shah R, Singhal S, Singh S, Piparva K, Katoch CDS. A systematic review and meta-analysis of tolerability, cardiac safety and efficacy of inclisiran for the therapy of hyperlipidemic patients. Expert Opin Drug Saf. 2024 Feb;23(2):187-198. doi: 10.1080/14740338.2023.2293201. Epub 2023 Dec 19. PMID 38063346
- [Derived] Raal FJ, Kallend D, Ray KK, Turner T, Koenig W, Wright RS, Wijngaard PLJ, Curcio D, Jaros MJ, Leiter LA, Kastelein JJP; ORION-9 Investigators. Inclisiran for the Treatment of Heterozygous Familial Hypercholesterolemia. N Engl J Med. 2020 Apr 16;382(16):1520-1530. doi: 10.1056/NEJMoa1913805. Epub 2020 Mar 18. PMID 32197277

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Inclisiran | Placebo
Started | 242 | 240
Completed | 235 | 231
Not Completed | 7 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Inclisiran | Placebo | Total
Number analyzed (Participants) | 242 | 240 | 482
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 189 | 185 | 374
  >=65 years | 53 | 55 | 108
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.4 (12.48) | 55.0 (11.81) | 54.7 (12.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 130 | 125 | 255
  Male | 112 | 115 | 227
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 8 | 15
  Not Hispanic or Latino | 235 | 232 | 467
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 7 | 5 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 8 | 7 | 15
  White | 226 | 227 | 453
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 12 | 11 | 23
  Netherlands | 19 | 19 | 38
  Sweden | 18 | 16 | 34
  United States | 33 | 32 | 65
  Czechia | 7 | 5 | 12
  Denmark | 23 | 26 | 49
  South Africa | 88 | 89 | 177
  Spain | 42 | 42 | 84

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in LDL-C From Baseline To Day 510
Time Frame: Baseline, Day 510
Population: ITT (intent-to-treat) Population
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Groups:
- Inclisiran: Inclisiran sodium 300 milligrams (mg) (equivalent to 284 mg inclisiran) administered as a subcutaneous injection on Day 1, Day 90, and then every 6 months.
- Placebo: Placebo administered as a subcutaneous injection of sterile saline solution (0.9% sodium chloride in water for injection) on Day 1, Day 90, and then every 6 months.
Arm/Group | Inclisiran | Placebo
Number analyzed (Participants) | 242 | 240
percent change | -41.15 [-44.52 to -37.77] | 8.37 [3.96 to 12.77]
Statistical Analysis 1: Comparison: Inclisiran vs Placebo; Test type: Superiority; p < .0001, ANCOVA — The a priori threshold for statistical significance was <0.05; Mean Difference (Final Values) = -49.52, 95% CI 2-sided [-55.04 to -43.99] — Represents the least squares mean difference from Placebo

2. Primary Outcome: Time-adjusted Percent Change in LDL-C From Baseline After Day 90 and up to Day 540
Description: Assessments performed at Baseline, Day 90, Day 540, time-adjusted percent change at Day 90 reported
Time Frame: Baseline, Day 90
Population: ITT (intent-to-treat) Population
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Inclisiran | Placebo
Number analyzed (Participants) | 242 | 240
percent change | -38.08 [-41.03 to -35.14] | 6.22 [3.26 to 9.17]
Statistical Analysis 1: Comparison: Inclisiran vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA — The a priori threshold for statistical significance was <0.05; Mean Difference (Final Values) = -44.30, 95% CI 2-sided [-48.48 to -40.12] — Represents the least squares mean difference from Placebo

3. Secondary Outcome: Absolute Change in LDL-C From Baseline to Day 510
Time Frame: Baseline, Day 510
Population: ITT (intent-to-treat) Population
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Inclisiran | Placebo
Number analyzed (Participants) | 242 | 240
mg/dL | -58.95 [-64.75 to -53.15] | 9.94 [4.10 to 15.78]
Statistical Analysis 1: Comparison: Inclisiran vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA — The a priori threshold for statistical significance was <0.05; Mean Difference (Final Values) = -68.89, 95% CI 2-sided [-77.11 to -60.67] — Represents the least squares mean difference from Placebo

4. Secondary Outcome: Time-adjusted Absolute Change in LDL-C From Baseline After Day 90 and up to Day 540
Description: Assessments performed at Baseline, Day 90, Day 540, absolute change at Day 90 reported
Time Frame: Baseline, Day 90
Population: ITT (intent-to-treat) Population
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Inclisiran | Placebo
Number analyzed (Participants) | 242 | 240
mg/dL | -56.58 [-60.98 to -52.17] | 6.17 [1.72 to 10.62]
Statistical Analysis 1: Comparison: Inclisiran vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA — The a priori threshold for statistical significance was <0.05; Mean Difference (Final Values) = -62.74, 95% CI 2-sided [-69.01 to -56.48] — Represents the least squares mean difference from Placebo

5. Secondary Outcome: Percentage Change in Proprotein Convertase Subtilisin/Kexin Type 9 (PCSK9) From Baseline to Day 510
Time Frame: Baseline, Day 510
Population: ITT (intent-to-treat) Population
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Inclisiran | Placebo
Number analyzed (Participants) | 242 | 240
percent change | -60.68 [-64.40 to -56.96] | 17.66 [13.91 to 21.42]
Statistical Analysis 1: Comparison: Inclisiran vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA — The a priori threshold for statistical significance was <0.05; Mean Difference (Final Values) = -78.34, 95% CI 2-sided [-83.65 to -73.04] — Represents the least squares mean difference from Placebo

6. Secondary Outcome: Percentage Change in Total Cholesterol From Baseline to Day 510
Time Frame: Baseline, Day 510
Population: ITT (intent-to-treat) Population
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Groups:
- Inclisiran: Inclisiran sodium 300 milligrams (mg) (equivalent to 284 mg inclisiran) administered as a subcutaneous injection on Day 1, Day 90, and then every 6 months.s.
Arm/Group | Inclisiran | Placebo
Number analyzed (Participants) | 242 | 240
percent change | -25.11 [-27.83 to -22.39] | 6.66 [3.96 to 9.36]
Statistical Analysis 1: Comparison: Inclisiran vs Placebo; Test type: Superiority — LS Mean Difference (95% CI) from Placebo; p < 0.0001, ANCOVA — The a priori threshold for statistical significance was <0.05; Mean Difference (Final Values) = -31.77, 95% CI 2-sided [-35.59 to -27.94] — Represents the least squares mean difference from Placebo

7. Secondary Outcome: Percent Change in Apolipoprotein B (Apo-B) From Baseline To Day 510
Time Frame: Baseline, Day 510
Population: ITT (intent-to-treat) Population
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Inclisiran | Placebo
Number analyzed (Participants) | 242 | 240
percent change | -33.14 [-35.91 to -30.36] | 2.93 [0.14 to 5.71]
Statistical Analysis 1: Comparison: Inclisiran vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA — The a priori threshold for statistical significance was <0.05; Mean Difference (Final Values) = -36.06, 95% CI 2-sided [-39.99 to -32.14] — Represents the least squares mean difference from Placebo

8. Secondary Outcome: Percent Change in Non-high-density Lipoprotein (HDL)-C From Baseline To Day 510
Time Frame: Baseline, Day 510
Population: ITT (intent-to-treat) Population
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Inclisiran | Placebo
Number analyzed (Participants) | 242 | 240
percent change | -34.93 [-38.46 to -31.40] | 7.43 [3.93 to 10.92]
Statistical Analysis 1: Comparison: Inclisiran vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA — The a priori threshold for statistical significance was <0.05; Mean Difference (Final Values) = -42.36, 95% CI 2-sided [-47.32 to -37.40] — Represents the least squares mean difference from Placebo

ADVERSE EVENTS:
Time Frame: Day 0 - 510
Description: The safety population for adverse event collection was 481 subjects which is different from the Intent-to-Treat (ITT) population used in efficacy analysis (482 subjects). One subject was randomized in the Inclisiran arm, but never received study drug, therefore this subject not included in the safety population.
Arm/Group | Inclisiran | Placebo
All-Cause Mortality (participants affected / at risk) | 1/241 | 1/240
Serious Adverse Events (participants affected / at risk) | 18/241 | 33/240
Other Adverse Events (participants affected / at risk) | 96/241 | 67/240
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Inclisiran (N=241) | Placebo (N=240)
Acute myocardial infarction (Cardiac disorders) | 2 | 1
Angina Pectoris (Cardiac disorders) | 1 | 0
Angina unstable (Cardiac disorders) | 1 | 4
Aortic valve stenosis (Cardiac disorders) | 2 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Cardiac failure acute (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 3
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Optic ischaemic neuropathy (Eye disorders) | 0 | 2
Gastritis erosive (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Hernia (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Biliary colic (Hepatobiliary disorders) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 1
Infective tenosynovitis (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1
Post procedural infection (Infections and infestations) | 0 | 1
Pyelitis (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 1
Tick-borne fever (Infections and infestations) | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1
Wound sepsis (Infections and infestations) | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haematuria (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Sensory disturbance (Nervous system disorders) | 0 | 1
Trigeminal neuralgia (Nervous system disorders) | 0 | 1
Device loosening (Product Issues) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 0 | 1
Major depression (Psychiatric disorders) | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Inclisiran (N=241) | Placebo (N=240)
Injection site reaction (General disorders) | 22 | 0
Influenza (Infections and infestations) | 13 | 21
Nasopharyngitis (Infections and infestations) | 28 | 20
Upper respiratory tract infection (Infections and infestations) | 16 | 16
Back pain (Musculoskeletal and connective tissue disorders) | 17 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-01-31): https://cdn.clinicaltrials.gov/large-docs/21/NCT03397121/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-13): https://cdn.clinicaltrials.gov/large-docs/21/NCT03397121/SAP_001.pdf